CLINICAL TRIAL: NCT05132049
Title: An Open-label, Randomized, Single-dose, 2-sequence, 2-period, Crossover Phase 1 Study to Evaluate the Pharmacokinetic Characteristics and the Safety After Administration of DA-5211 and Co-administration of DA-5211-R1 and DA-5211-R2 in Healthy Adult Volunteer
Brief Title: Pharmacokinetics and Safety Profiles After Administration of DA-5211 and Co-administration of DA-5211-R1 and DA-5211-R2 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DA5211_BE_I
Record Dates: First submitted 2021-11-16; First posted 2021-11-23 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental)
  Interventions: Drug: DA-5211; Drug: DA-5211-R1 + DA-5211-R2
- Sequence B (Experimental)
  Interventions: Drug: DA-5211; Drug: DA-5211-R1 + DA-5211-R2

INTERVENTIONS:
Drug: DA-5211 — single dose administration (DA-5211 one tablet once a day)
Drug: DA-5211-R1 + DA-5211-R2 — single dose administration (DA-5211-R1 one tablet once a day + DA-5211-R2 one tablet once a day)

SUMMARY:
Pharmacokinetics and safety Profiles after administration of DA-5211 and co-administration of DA-5211-R1 and DA-5211-R2 in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* BMI between 18 and 30 kg/m2
* Body weight: Male≥50kg, Female≥45kg
* Subjects who have signed an informed consent themselves after receiving detailed explanation about clinical study

Exclusion Criteria:

* Subjects with allergy or drug hypersensitivity
* Subjects with clinically significant medical history
* Subjects with history of drug abuse or addicted

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-12-18 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
AUCt | pre-dose~72 hours post-dose
  area under the curve
Cmax | pre-dose~72 hours post-dose
  maximum plasma concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Bumin Hospital, Seoul, South Korea